CLINICAL TRIAL: NCT05049395
Title: HFNO Reducing the Incidence of Hypoxia During the Procedure of Hysteroscopy Sedated With Propofol，a Randomized, Controlled Trial
Brief Title: HFNO Reducing the Incidence of Hypoxia for Hysteroscopy Sedated With Propofol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RJ20210904
Record Dates: First submitted 2021-07-13; First posted 2021-09-20 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Endometritis; Tuberculous Endometritis; Subseptate Uterus; Endometrial Polyps
Keywords: HFNO; Hysteroscopy; Sedation; Hypoxia
MeSH Terms: conditions — Endometritis; Septate Uterus; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The patients are administered oxygen of 3L-6L/min until the end of the hysteroscopy operation.
  Interventions: Device: Regular oxygen
- HFNO group (Experimental): The patients are administered oxygen of 30L-60L/min until the end of the hysteroscopy operation.
  Interventions: Device: High Flow Nasal Cannula oxygen (HFNO)

INTERVENTIONS:
Device: High Flow Nasal Cannula oxygen (HFNO) — The AIRVO2 is set at 30L/min, FiO2 100%, and 37℃ before anesthesia induction，and then 60L/min until the end of the procedure of sedated hysteroscopy.
  Arms: HFNO group
Device: Regular oxygen — The patients are administered oxygen of 3L-6L/min until the end of the hysteroscopy operation.
  Arms: Control group

SUMMARY:
To determine whether high-flow nasal cannula oxygen can reduce the incidence of hypoxia during the procedure of sedated hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old ≤ age ≤ 50 years old, female.
2. Undergoing hysteroscopy sedated with propofol for diagnosis or treatment.
3. Informed consent
4. BMI≤28kg/m2.
5. ASA physical status Ⅰ~ Ⅱ.

Exclusion Criteria:

1. Epistaxis, nasal congestion and nasal mucosal damage.
2. Confirmed brain disease (cranial trauma, tumor, stroke, cognitive dysfunction etc.).
3. Confirmed severe heart disease (heart failure, angina pectoris, myocardial infarction, arrhythmia, etc.).
4. Confirmed severe lung diseases (upper respiratory tract infection, asthma, bronchitis, COPD, bullae, pulmonary embolism, pulmonary edema, lung cancer, etc.).
5. Pregnant women.
6. Acute and chronic hepatitis or liver cirrhosis with severe abnormal liver function.
7. Acute and chronic nephritis with severe abnormal renal function or renal failure.
8. Needing oxygen inhalation for underlying diseases.
9. Emergency surgery.
10. Combined with multiple trauma.
11. Allergic to soybean

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 960 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  75%≤SpO2<90% and <60S

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90%≤SpO2<95%

OTHER OUTCOMES:
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 <90% for >= 60 s
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Overall Officials: Su Diansan, PhD, Principal Investigator — Department of Anesthesiology
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China